CLINICAL TRIAL: NCT02657356
Title: A Study of the Efficacy and Safety of Bardoxolone Methyl in Patients With Connective Tissue Disease-associated Pulmonary Arterial Hypertension
Brief Title: Bardoxolone Methyl in Patients With Connective Tissue Disease-associated Pulmonary Arterial Hypertension - CATALYST
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Exposure of these high-risk patients to clinic or in-person visits during the pandemic presented an unacceptable risk to their health
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RTA 402-C-1504
Record Dates: First submitted 2016-01-13; First posted 2016-01-15 (Estimated); Results first posted 2023-05-19 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Connective Tissue Disease-Associated Pulmonary Arterial Hypertension
Keywords: Pulmonary Hypertension; Pulmonary Arterial Hypertension; Connective Tissue Disease-Associated Pulmonary Arterial Hypertension; Bardoxolone methyl; PAH; RTA 402; 6-minute walk distance
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — bardoxolone methyl; ORF 50 transactivator

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo capsules (Placebo Comparator): Placebo capsules will be administered orally once a day for 24 weeks.
  Interventions: Drug: Placebo capsules
- Bardoxolone methyl capsules (Experimental): Each patient will receive bardoxolone methyl capsules administered orally once a day for 24 weeks. Starting dosage for each patient is 5 mg and will dose-escalate to 10 mg at Week 4, unless contraindicated clinically.
  Interventions: Drug: Bardoxolone methyl capsules

INTERVENTIONS:
Drug: Placebo capsules
  Arms: Placebo capsules
Drug: Bardoxolone methyl capsules
  Other Names: RTA 402 capsules
  Arms: Bardoxolone methyl capsules

SUMMARY:
This study assesses the safety and efficacy of bardoxolone methyl relative to placebo in patients with connective tissue disease-associated pulmonary arterial hypertension to determine the recommended dose range and evaluate the change from baseline in 6-minute walk distance (6MWD) following 24 weeks of study participation.

DETAILED DESCRIPTION:
This double-blind, randomized, placebo-controlled trial will study the safety, tolerability, and efficacy of bardoxolone methyl in qualified patients with World Health Organization Group I Connective Tissue Disease Pulmonary Arterial Hypertension (WHO Group I CTD-PAH).

Qualified patients will be randomized 1:1 to either bardoxolone methyl or placebo to be administered once daily for 24 weeks. Patients randomized to placebo will remain on placebo throughout the study. Patients randomized to bardoxolone methyl will start at 5 mg and will dose-escalate to 10 mg at Week 4 unless contraindicated clinically. Dose de-escalation is permitted during the study if indicated clinically.

All patients in the study will follow the same visit and assessment schedule. Following randomization, patients will be scheduled to be assessed in person during treatment at Weeks 1, 2, 4, 6, 8, 16, and 24 and by telephone contact on Days 3, 10, 21, 31, 38, 84, and 140. Patients will also be scheduled to be assessed at an in person follow up visit at Week 28, four weeks after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 18.5 kg/m2;
* Symptomatic pulmonary hypertension WHO/NYHA FC class II and III;
* WHO Group I PAH associated with connective tissue disease;
* Had a diagnostic right heart catheterization performed and documented within 36 months prior to Day 1 that confirmed a diagnosis of PAH according to all the following criteria:

  * Mean pulmonary artery pressure ≥ 25 mm Hg (at rest);
  * Pulmonary capillary wedge pressure (PCWP) ≤ 15 mm Hg;
  * Pulmonary vascular resistance > 240 dyn.sec/cm5 or > 3 mm Hg/liter (L)/minute;
* Has BNP level ≤ 400 pg/mL;
* Had an average 6MWD ≥ 150 meters on two consecutive tests performed on different days prior to randomization, with both tests measuring within 15% of one another;
* Has been receiving no more than two (2) approved disease-specific PAH therapies. PAH therapy must have been at a stable dose for at least 90 days prior to Day 1. No additions or changes should be made to PAH therapies and doses should remain stable for the duration of the study;
* Has maintained a stable dose for 30 days prior to Day 1 if receiving any of the following therapies that may affect PAH: vasodilators (including calcium channel blockers), digoxin, L-arginine supplementation, or oxygen supplementation. No additions or changes should be made to therapies and doses should remain stable for the duration of the study;
* If receiving treatment for CTD with prednisone or any other drugs, doses must remain stable for at least 30 days prior to Day 1 and for the duration of the study Had pulmonary function tests (PFTs) within 90 days prior to Day 1 with total lung capacity ≥ 65% (predicted);
* Had a ventilation-perfusion (V/Q) lung scan, spiral/helical/electron beam computed tomography (CT), or pulmonary angiogram prior to Day 1 that shows no evidence of thromboembolic disease (i.e., should note normal or low probability for pulmonary embolism). If V/Q scan was abnormal (i.e., results other than normal or low probability), then a confirmatory CT or selective pulmonary angiography must exclude chronic thromboembolic pulmonary hypertension;
* Has adequate kidney function defined as an estimated glomerular filtration rate (eGFR) ≥ 45 mL/min/1.73 m2 as measured by the central lab;
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures;
* Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study prior to initiation of any patient-mandated procedures

Exclusion Criteria:

* Participation in other investigational clinical studies involving interventional products being tested or used in a way different from the approved form or when used for an unapproved indication within 30 days prior to Day 1;
* Initiation of an exercise program for cardio-pulmonary rehabilitation within 90 days prior to Day 1 or planned initiation during the study;
* Stopped receiving any PAH chronic therapy within 60 days prior to Day 1;
* Received a dose of prednisone > 20 mg/day (or equivalent dose if other corticosteroid) within 30 days prior to Day 1;
* Received intravenous (iv) or subcutaneous (sc) prostacyclin/prostacyclin analogues within 90 days prior to Day 1;
* Received intravenous inotropes within 30 days prior to Day 1;
* Has uncontrolled systemic hypertension as evidenced by sitting systolic blood pressure (BP) > 160 mm Hg or sitting diastolic BP > 100 mm Hg during Screening after a period of rest;
* Has systolic BP < 90 mm Hg during Screening after a period of rest;
* Has a history of clinically significant left-sided heart disease and/or clinically significant cardiac disease, including but not limited to any of the following:

  * Congenital or acquired valvular disease if clinically significant apart from tricuspid valvular insufficiency due to pulmonary hypertension;
  * Pericardial constriction;
  * Restrictive or congestive cardiomyopathy;
  * Left ventricular ejection fraction < 40% per echocardiogram (ECHO) within 90 days of Day 1;
  * Symptomatic coronary artery disease within the last 3 years;
* Acutely decompensated heart failure within 30 days prior to Day 1, per investigator assessment;
* Has more than two of the following clinical risk factors for left ventricular diastolic dysfunction:

  * Age > 65 years;
  * BMI ≥ 30 kg/m2;
  * History of systemic hypertension;
  * History of type 2 diabetes;
  * History of atrial fibrillation;
  * History of atrial septostomy within 180 days prior to Day 1;
  * History of uncontrolled obstructive sleep apnea;
* Has a history of portal hypertension or chronic liver disease, including hepatitis B and/or hepatitis C (with evidence of recent infection and/or active virus replication) defined as mild to severe hepatic impairment (Child-Pugh Class A-C);
* Serum aminotransferase (ALT or AST) levels > 1.5X the upper limit of normal (ULN) at Screening;
* Hemoglobin (Hgb) concentration < 8.5 g/dL at Screening;
* Diagnosis of Down syndrome;
* History of malignancy within 5 years prior to screening, with the exception of localized skin or cervical carcinomas;
* Untreated or uncontrolled active bacterial, fungal, or viral infection;
* Known or suspected active drug or alcohol abuse, per investigator judgment;
* Use of Herbalife supplements within 14 days prior to Day 1;
* Major surgery within 30 days prior to Day 1 or planned to occur during the course of the study;
* Unwilling to practice acceptable methods of birth control (both males who have partners of childbearing potential and females of childbearing potential) during screening, while taking study drug, and for at least 30 days after the last dose of study drug is ingested;
* Use of inhaled nitric oxide within 7 days prior to Screening and Day 1 visits, excluding acute vasodilator testing during diagnostic cardiac catheterization;
* Women who are pregnant or breastfeeding;
* Any disability or impairment that would prohibit performance of the 6MWT;
* Any abnormal laboratory level that, in the opinion of the investigator, would put the patient at risk by trial enrollment;
* Patient is, in the opinion of the investigator, unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason;
* Known hypersensitivity to any component of the study drug;
* Unable to communicate or cooperate with the investigator because of language problems, poor mental development, or impaired cerebral function.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (106):
- United States (37):
  - Banner University Medical Center, Phoenix Advanced Lung Disease Institute, Phoenix, Arizona
  - Arizona Pulmonary Specialists, Phoenix, Arizona
  - Cedars Sinai Medical Center, Beverly Hills, California
  - Regents of The University of California, Fresno, California
  - University of California San Diego, La Jolla, California
  - David Geffen School of Medicine UCLA, Los Angeles, California
  - Pacific Pulmonary Research, Inc., San Diego, California
  - Santa Barbara Pulmonary Associates, Santa Barbara, California
  - Harbor - UCLA Medical Center, Torrance, California
  - Georgetown University Medical Center - Department of Rheumatology, Washington D.C., District of Columbia
  - University of Miami Miller School of Medicine, Miami, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Augusta University, Augusta, Georgia
  - Piedmont-Georgia Lung, Austell, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of New Mexico, Albuquerque, New Mexico
  - NYU Langone Health, New York, New York
  - University of Rochester - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Wexner Medical Center at The Ohio State University, Columbus, Ohio
  - Integris Nazih Zuhdi Transplant Institute, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
- Argentina (9):
  - Fundación Favaloro, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Hospital Británico de Buenos Aires, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Centro Médico Dra de Salvo, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Instituto de Investigaciones Clínicas Mar Del Plata, Buenos Aires, Mar Del Plata
  - Instituto De Enfermedades Respiratorias E Investigacion Medica, Buenos Aires, Villa Vatteone
  - Instituto de Cardiologia de Corrientes Juana Francisca Cabral, Corrientes
  - Hospital Cordoba, Córdoba
  - Hospital Privado Centro Médico de Córdoba, Córdoba
  - Hospital de Alta Complejidad "Pte. J. D. Perón", Formosa
- Australia (5):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
- Belgium (2):
  - UZ Leuven, Leuven, Vlaams Brabant
  - Hôpital Erasme, Brussels
- Brazil (5):
  - Hospital de Messejana, Fortaleza, Ceará
  - Irmandade Da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Dia do Pulmão, Blumenau, Santa Catarina
  - Hospital São Paulo, São Paulo
  - Instituto do Coração - HCFMUSP, São Paulo
- Canada (5):
  - Peter Lougheed Centre, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
  - Centre Hospitalier de l'Université Laval, Sainte-Foy, Quebec
- Czechia (2):
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Institut klinicke a experimentalni mediciny, Prague
- Germany (8):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitatsklinkum Erlangen, Erlangen, Bavaria
  - Universität Greifswald, Greifswald, Mecklenburg-Vorpommern
  - DRK Kliniken Berlin Westend, Berlin
  - Universitätsklinikum Köln, Cologne
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - Thorax Klinik, Heidelberg
- Israel (2):
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Rabin Medical Center, Petah Tikva
- Japan (12):
  - Nippon Medical School Hospital, Tokyo, Bunkyo-ku
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - National Hospital Organization Okayama Medical Center, Okayama, Okayama-ken
  - Chiba University Hospital, Chiba
  - Gunma University School of Medicine, Gunma
  - Kobe University Hospital, Kobe
  - Nagoya Medical Center, Nagoya
  - Hokkaido University Hospital, Sapporo
  - Kurume University Medical Center, Sendai
  - National Cerebral and Cardiovascular Center, Suita
  - Fujita Health University Hospital, Toyoake
- Mexico (5):
  - Hospital Civil Fray Antonio Alcalde, Guadalajara, Jalisco
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico City
  - Instituto Nacional de Cardiologia Dr. Ignacio Chavez, Mexico City, Mexico City
  - Hospital Universitario Dr. Jose Eleuterio González, Monterrey, Nuevo León
  - Unidad de Investigación Clínica En Medicina SC, Monterrey, Nuevo León
- Vrije Universiteit Amsterdam, Amsterdam, North Holland, Netherlands
- Philippines (5):
  - Angeles University Foundation Medical Center (AUFMC), Angeles City
  - Mary Mediatrix Medical Center (MMMC), Lipa
  - Makati Medical Center (MMC), Makati
  - Philippine General Hospital (PGH), Manila
  - Philippine Heart Center (PHC), Quezon City
- Spain (6):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Hospital Virgen de La Salud, Toledo
- United Kingdom (2):
  - Golden Jubilee National Hospital, Glasgow
  - Royal Free Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Capsules: Placebo capsules administered orally once a day for 24 weeks with sham titration.
- Bardoxolone Methyl Capsules: Bardoxolone methyl capsules administered orally once a day for 24 weeks. Starting dosage for each patient was 5 mg and dose-escalated to 10 mg at Week 4, unless contraindicated clinically.
Period: Overall Study
Arm/Group | Placebo Capsules | Bardoxolone Methyl Capsules
Started | 102 | 100
Completed | 82 | 85
Not Completed | 20 | 15
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Terminated by Sponsor | 8 | 5
Not completed — Rolled over to EAP study | 6 | 4

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population (all randomized patients categorized by their assigned treatment group regardless of treatment exposure)
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Capsules | Bardoxolone Methyl Capsules | Total
Number analyzed (Participants) | 102 | 100 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (13.17) | 55 (13.57) | 55.7 (13.36)
Age, Customized [Median (Full Range); unit: years]
  Median Age | 60 [21 to 75] | 57 [29 to 75] | 59 [21 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 88 | 179
  Male | 11 | 12 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 27 | 59
  Not Hispanic or Latino | 70 | 73 | 143
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 16 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 6 | 16
  White | 78 | 76 | 154
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  Argentina | 14 | 12 | 26
  Australia | 8 | 7 | 15
  Belgium | 2 | 1 | 3
  Brazil | 5 | 4 | 9
  Canada | 5 | 5 | 10
  Czechia | 1 | 2 | 3
  Germany | 1 | 5 | 6
  Spain | 5 | 3 | 8
  United Kingdom | 1 | 2 | 3
  Israel | 2 | 2 | 4
  Japan | 7 | 9 | 16
  Mexico | 4 | 8 | 12
  Netherlands | 1 | 1 | 2
  Philippines | 1 | 4 | 5
  United States | 45 | 35 | 80
Six Minute Walk Distance (6MWD) [Mean (Standard Deviation); unit: meters] — Baseline 6MWD measured using the Six Minute Walk Test (6MWT)
  meters | 380.4 (91.19) | 389.1 (107.78) | 384.7 (99.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Six-minute-walk Distance (6MWD) Relative to Placebo at Week 24
Time Frame: Baseline through 24 weeks after participant receives the first dose
Population: ITT population (all randomized patients categorized by their assigned treatment group regardless of treatment exposure)
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | Placebo Capsules | Bardoxolone Methyl Capsules
Number analyzed (Participants) | 102 | 100
meters | 9.25 (4.954) | -3.61 (4.952)
Statistical Analysis 1: Comparison: Placebo Capsules vs Bardoxolone Methyl Capsules; Test type: Superiority; p = 0.0683, Mixed Models Analysis; Covariates: screening 6MWT, day 1 hemoglobin, treatment grp, # of PAH medications, time, interactions btwn treatment & time, and screening 6MWT & time; LS Mean difference (Net) = -12.86, 95% CI 2-sided [-26.69 to 0.98], Standard Error of Mean 7.012 — Difference is bardoxolone methyl - placebo

2. Secondary Outcome: Time to First Persistent Clinical Improvement Event
Description: At least one of the following four criteria must have been met:
  1. Improvement by at least one WHO functional class coupled with no more than a 15% decrease from baseline in 6MWT
  2. Increase from baseline in 6MWT by at least 10% and stability or improvement in the WHO functional class
  3. Decrease from baseline in creatine kinase (a surrogate biomarker for muscle injury and inflammation) by at least 10% and no worsening in WHO functional class and no more than a 15% decrease from baseline in 6MWT
  4. Improvement in estimated glomerular filtration rate eGFR ≥10% of baseline The persistence of the change in WHO functional class, 6MWT, eGFR, or creatine kinase must be confirmed by a subsequent assessment at least 14 days after the initial assessment, or at the next scheduled assessment. If persistent improvement is confirmed, the date of the event was considered the initial assessment of improved WHO functional class, 6MWT, eGFR, or creatine kinase.
Time Frame: Baseline through the end of the study
Population: ITT population (all randomized patients categorized by their assigned treatment group regardless of treatment exposure)
Measure: Mean (Standard Error); unit: weeks
Arm/Group | Placebo Capsules | Bardoxolone Methyl Capsules
Number analyzed (Participants) | 102 | 100
weeks | 17.9 (1.263) | 6.62 (0.646)
Statistical Analysis 1: Comparison: Placebo Capsules vs Bardoxolone Methyl Capsules; Test type: Superiority; p = 0.0004, Chi-squared; Hazard Ratio (HR) = 1.984, 95% CI 2-sided [1.360 to 2.895] — Estimated from Cox Regression adjusted by baseline PAH medication status (0-1 vs 2) as the covariate. Hazard ratio >1 indicates a beneficial effect that favors bardoxolone methyl

ADVERSE EVENTS:
Time Frame: 28 weeks
Description: All adverse events that are observed or reported by the patient during the study (from the time of administration of the first dose at Day 1 until the final visit) must be reported, regardless of their relationship to study drug or their clinical significance.
Arm/Group | Placebo Capsules | Bardoxolone Methyl Capsules
All-Cause Mortality (participants affected / at risk) | 1/102 | 0/100
Serious Adverse Events (participants affected / at risk) | 18/102 | 16/100
Other Adverse Events (participants affected / at risk) | 79/102 | 85/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Capsules (N=102) | Bardoxolone Methyl Capsules (N=100)
Arteriospasm coronary (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Capsules (N=102) | Bardoxolone Methyl Capsules (N=100)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 6 (6)
Palpitations (Cardiac disorders) | 2 (2) | 3 (3)
Dry eye (Eye disorders) | 3 (3) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 3 (3)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 6 (6) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 21 (25) | 13 (15)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastritis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 9 (10)
Nausea (Gastrointestinal disorders) | 11 (13) | 12 (12)
Vomiting (Gastrointestinal disorders) | 7 (8) | 8 (8)
Fatigue (General disorders) | 13 (13) | 9 (9)
Non-cardiac chest pain (General disorders) | 6 (7) | 3 (3)
Oedema peripheral (General disorders) | 12 (14) | 9 (9)
Pyrexia (General disorders) | 3 (3) | 3 (3)
Bronchitis (Infections and infestations) | 5 (5) | 7 (7)
Gastroenteritis (Infections and infestations) | 2 (2) | 4 (4)
Influenza (Infections and infestations) | 7 (7) | 2 (2)
Nasopharyngitis (Infections and infestations) | 5 (5) | 11 (13)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Sinusitis (Infections and infestations) | 4 (4) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 11 (15) | 19 (27)
Urinary tract infection (Infections and infestations) | 6 (11) | 8 (11)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 6 (6)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 6 (6)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 5 (5)
Brain natriuretic peptide increased (Investigations) | 2 (2) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 8 (8)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 1 (1) | 5 (5)
Weight decreased (Investigations) | 2 (2) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 9 (9)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 4 (6)
Gout (Metabolism and nutrition disorders) | 0 (0) | 5 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (13) | 3 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 9 (10)
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (7) | 17 (19)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (9)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1)
Dizziness (Nervous system disorders) | 12 (12) | 8 (10)
Dizziness postural (Nervous system disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 21 (28) | 14 (15)
Presyncope (Nervous system disorders) | 1 (1) | 3 (4)
Depression (Psychiatric disorders) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 6 (6) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 9 (9)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2016-10-18): https://cdn.clinicaltrials.gov/large-docs/56/NCT02657356/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/56/NCT02657356/SAP_001.pdf